CLINICAL TRIAL: NCT06546306
Title: Efficacy and Safety of the Touch® Dual Mobility Trapeziometacarpal Prosthesis and Its Surgical Instruments Set in the Treatment of Basal Thumb Osteoarthritis: Post-market Observational Clinical Study.
Brief Title: Post Market Clinical Follow-Up TOUCH® CMC 1
Status: Active, not recruiting | Type: Observational
Sponsor: Keri Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-A02352-55
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis Thumb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: TOUCH® CMC 1 — TOUCH® prosthesis is a total CMC 1 (1st Carpo-metacarpal) joint replacement prosthesis.

SUMMARY:
Because severe pain, weakened pinch and grip strength produce functional disabilities, the basal joint of the thumb is the most common site of surgical reconstruction in the upper limb due to OA.

The cement-free dual mobility Touch® prosthesis consists of a metacarpal implant (stem), a trapezium implant (cup), and a connection implant (neck).

The main objective of this study is to describe the performance and safety of the Touch® prosthesis used with its instruments set in accordance with its intention and CE marking in force.

Performance and safety will be assessed over the short and long term in accordance with the life cycle of the Touch® prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years),
* Patients suffering from rhizarthrosis (I - IV based on the Dell classification),
* Pain >3 on the VAS scale,
* Patients to undergo a replacement of the trapeziometacarpal joint with the Touch® dual mobility trapeziometacarpal prosthesis.

Exclusion Criteria:

* Pregnant women,
* Patients with contraindications to surgery in general,
* Patients suffering from Temporary Regional Pain Syndrome (TRPS),
* Patients with a severe or chronic, local or systemic infection,
* Patients with severe muscle, neurological or vascular impairments affecting the trapezium-metacarpal joint,
* Patients with bone demineralization or destruction that may affect the proper fixation of the implant,
* Patients whose bone dimensions are incompatible with the implant dimensions,
* The combination of the Touch® prosthesis with other components of another origin is not authorized,
* Patients with allergies to the components of the product or with known allergies (chromium, cobalt, nickel),
* Patients with an intellectual disability who cannot, therefore, follow the instructions of their surgeon,
* Patient with scaphoid-trapezium-trapezoid (STT) arthritis,
* Patient requiring revision of a trapeziometacarpal prosthesis,
* Patient who has undergone a TMC joint infiltration within 3 months of the expected date of replacement of the joint with a Touch® prosthesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any type of population requiring a surgical procedure covered by the device indications and contraindications.
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Mobility and pain | 3 months
  At 3 months post-surgery, the proportion of patients with a Kapandji score > 8 and a pain score ≤ 3 on a VAS scale.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre de la main du Pays d'Aix, Aix-en-Provence
  - Clinic of Chataigneraie, Beaumont
  - Orthopaedics and Trauma Surgery Practice, Bezannes
  - Médipôle De Savoie, Challes-les-Eaux
  - Medical Office of Dr TCHURUKDICHIAN, Dijon
  - Medical Office Archimed, Lesquin

IPD SHARING:
Plan to Share IPD: No